CLINICAL TRIAL: NCT01326208
Title: Influence of Different Strategies to Optimize Positive End-expiratory Pressure on Pulmonary Gas Exchange, Perfusion/Ventilation Matching and Homogeneity of Ventilation in Patients With Acute Lung Injury
Brief Title: Strategies to Optimize Positive End-expiratory Pressure (PEEP) in Patients With Acute Lung Injury
Acronym: EIT-PEEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Prof. Dr. Christian Putensen, University of Bonn, Dep. of Anesthesiology and Intensive Care Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EIT-PEEP-2010
Record Dates: First submitted 2010-07-15; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Respiratory Failure
Keywords: electrical impedance tomography; positive end-expiratory pressure; regional ventilation delay index
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute Lung Injury / ARDS (Experimental): Patient under mechanical suffering from ALI or ARDS
  Interventions: Procedure: PEEP titration

INTERVENTIONS:
Procedure: PEEP titration — PEEP is set according to the following protocols, respectively, in a randomized order: ARDSnet table, Open Lung strategy, guided by EIT
  Other Names: electrical impedance tomography guided setting of PEEP

SUMMARY:
The purpose of this study in patients suffering from acute lung injury is to determine whether positive end-expiratory pressure (PEEP) setting guided by electrical impedance tomography (EIT) influences pulmonary gas exchange, lung mechanics, ventilation/perfusion matching and homogeneity of regional ventilation when compared to other PEEP setting strategies such as the open lung concept or the ARDSnet protocol.

ELIGIBILITY:
Inclusion Criteria:

* acute lung injury, need for optimization of ventilatory settings

Exclusion Criteria:

* preexisting chronical lung disease, pneumothorax, pace maker, hemodynamical instability, increased intracranial pressure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
homogeneity of regional ventilation delay | up to eight hours
  influence of different PEEP titration strategies on homogeneity of regional ventilation delay measured by electrical impedance tomography

SECONDARY OUTCOMES:
pulmonary gas exchange, lung mechanics and ventilation/perfusion matching | up to eight hours
  influence of different PEEP titration strategies on pulmonary gas exchange, lung mechanics and ventilation/perfusion matching

CONTACTS AND LOCATIONS:
Overall Officials: Christian Putensen, MD, Prof, Study Chair — University of Bonn; Thomas Muders, MD, Principal Investigator — University of Bonn
Locations (1):
- University Hospital, Bonn, Germany